CLINICAL TRIAL: NCT03567863
Title: Multicentric Randomized Study Comparing the Histological and Molecular Material Quality Obtained by EUS-FNB of Pancreatic Mass With Two "Biopsic" Needles: the 20-gauge Procore® (Cook) and the 22-gauge Acquire® (Boston Scientific)
Brief Title: Study Comparing Pancreatic EUS-FNB With the 20-gauge Procore® and the 22-gauge Acquire® Needles
Acronym: HISTOPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, MD, Principal Investigator, Société Française d'Endoscopie Digestive
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018-A00276-49
Record Dates: First submitted 2018-05-29; First posted 2018-06-26 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Pancreas Cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: the order of use of the 2 needles is not communicated to the cytologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): The two punctures performed successively with the 20-GAUGE PROCORE® (COOK) and the 22-GAUGE ACQUIRE® (BOSTON SCIENTIFIC)
  20-GAUGE PROCORE® first, then 22-GAUGE ACQUIRE®
  Interventions: Device: 20-GAUGE PROCORE® first, then 22-GAUGE ACQUIRE®
- Group B (Active Comparator): The two punctures performed successively with the 22-GAUGE ACQUIRE® (BOSTON SCIENTIFIC) and the 20-GAUGE PROCORE® (COOK)
  22-GAUGE ACQUIRE® first, then 20-GAUGE PROCORE®
  Interventions: Device: 22-GAUGE ACQUIRE® first, then 20-GAUGE PROCORE®

INTERVENTIONS:
Device: 20-GAUGE PROCORE® first, then 22-GAUGE ACQUIRE® — The two punctures performed successively with the 20-GAUGE PROCORE® (COOK) and the 22-GAUGE ACQUIRE® (BOSTON SCIENTIFIC)
  Arms: Group A
Device: 22-GAUGE ACQUIRE® first, then 20-GAUGE PROCORE® — The two punctures performed successively with the 22-GAUGE ACQUIRE® (BOSTON SCIENTIFIC) and the 20-GAUGE PROCORE® (COOK)
  Arms: Group B

SUMMARY:
Multicenter randomized prospective study

Criteria for inclusion:

Patients admitted for EUS-FNB of a pancreatic mass

Goals of the study:

To compare the results of blinded punctures for suspicion of pancreatic tumor performed under endoscopic ultrasound in our center (Digestive Endoscopy Unit of the Digestive Pole Paris Bercy, PDPB), in terms of diagnosis and quality of histopathological material obtained with the help of 20G Procore, Cook and 22G Acquire needles, Boston Scientific.

Main criterion:

- Biopsy core length of target tissue obtained by needle pass

Number of patients:

60 patients

Duration of the study:

1 year

DETAILED DESCRIPTION:
Type of study:

Multicenter randomized prospective study

Criteria for inclusion:

Patients admitted for ENDOSCOPIC ULTRASOUND FINE NEEDLE BIOPSY (EUS-FNB) of a pancreatic mass

Exclusion criteria:

Patients with an extra-pancreatic mass puncture Echendoscopic puncture contraindication or vascular interposition

Goals of the study:

To compare the results of blinded punctures for suspicion of pancreatic tumor performed under endoscopic ultrasound in our center (Digestive Endoscopy Unit of the Digestive Pole Paris Bercy, PDPB), in terms of diagnosis and quality of histopathological material obtained with the help of 20G Procore, Cook and 22G Acquire needles, Boston Scientific.

Evaluation criteria :

Main criterion:

- Biopsy core length of target tissue obtained by needle pass

Secondary criteria

* Presence of a core biopsy specimen
* Sensitivity of EUS-FNB for the diagnosis of adenocarcinoma of the pancreas
* False negative rate, Negative predictive value for the diagnosis of pancreatic adenocarcinoma
* Computer Aided Morphometric Evaluation of the Tumor + Stroma Surface on All core biopsy specimens
* Success rate of isolation of tumor cells and determination of transcriptomic signatures of pancreatic adenocarcinoma subtypes
* Immediate complications of puncture
* Variation in the quality of the puncture following the trans-duodenal or trans-gastric access route
* Technical failure rate of puncture
* Optional: inter and intra-observer evaluation of the anatomopathological criteria used (presence of a biopsy core, length of target tissue core per needle passage)

Number of patients:

60 patients

Duration of the study:

1 year

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to one of the investigative centers for endoscopic pancreatic puncture during the period from April 1, 2018 to April 1, 2019
* Patient whose age is greater than or equal to 18 years and less than 90 years
* Patient ASA 1, ASA 2, ASA 3 (ASA: American Society of Anaesthesiologists Classification)
* Lack of participation in another clinical study
* Signed informed consent

Exclusion Criteria:

* Patients punctured with an extra-pancreatic mass
* Patient under the age of 18 or over 90
* Patient ASA 4, ASA 5
* Pregnant woman
* Patient with coagulation abnormalities preventing puncture: TP <50%, Platelets <50000 / mm3, effective anticoagulation in progress, clopidogrel in progress
* Vascular or ductal or surgical fixation (Billroth II, Roux in Y) preventing endoscopic access to the lesion to be punctured
* Patient unable to personally consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-24 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
cumulative length of tissue core biopsies per needle pass | in the 7 days after procedure
  cumulative length of tissue core biopsies per needle pass in mm

SECONDARY OUTCOMES:
Presence of core biopsy specimen | in the 7 days after procedure
  Presence of core biopsy specimen
Sensitivity | in the 7 days or 6 months
  EUS-FNB Sensitivity for the diagnosis of adenocarcinoma of the pancreas
Specificity | in the 7 days or 6 months
  EUS-FNB Specificity for the diagnosis of adenocarcinoma of the pancreas
Positive Predictive Value | in the 7 days or 6 months
  EUS-FNB Positive predictive value for the diagnosis of adenocarcinoma of the pancreas
Negative Predictive Value | in the 7 days or 6 months
  EUS-FNB Negative Predictive Value for the diagnosis of adenocarcinoma of the pancreas
Computer Aided Morphometric Evaluation of the Tumor + Stroma Surface | 6 months
  Computer Aided Morphometric Evaluation of the Tumor + Stroma Surface on All Core biopsies
Success rate of isolation of tumor cells | 6 months
  Success rate of isolation of tumor cells
Morbidity | 7 days
  Puncture Morbidity (acute pancreatitis, haemorrhage)
Feasibility | during procedure
  Technical failure rate of puncture because of a impossibility to access to pancreatic mass with the needle (due to the needle stiffness)
inter evaluation of the anatomopathological criteria used (presence of a biopsy core, length of target tissue core per needle pass) | 7 days
  inter evaluation of the anatomopathological criteria used (presence of a biopsy core, length of target tissue core per needle pass)
determination of transcriptomic signatures of pancreatic adenocarcinoma subtypes | 6 months
  determination of transcriptomic signatures of pancreatic adenocarcinoma subtypes
intra-observer evaluation of the anatomopathological criteria used | 7 days
  intra-observer evaluation of the anatomopathological criteria used

CONTACTS AND LOCATIONS:
Overall Officials: David Karsenti, MD, Principal Investigator — Société Française d'Endoscopie Digestive
Locations (1):
- David Karsenti, Charenton-le-Pont, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen TY, Cao JW, Jin C, Ji Y, Zhong L, Wang LM, Cui N, Di Y, Bao Y, Zhong N, Zhang YQ, Zhou PH. Comparison of specimen quality among the standard suction, slow-pull, and wet suction techniques for EUS-FNA: A multicenter, prospective, randomized controlled trial. Endosc Ultrasound. 2022 Sep-Oct;11(5):393-400. doi: 10.4103/EUS-D-21-00163. PMID 36255027
- [Derived] Ishikawa H, Yamada M, Sato Y, Tanaka S, Akiko C, Tajika M, Doyama H, Takayama T, Ohda Y, Horimatsu T, Sano Y, Tanakaya K, Ikematsu H, Saida Y, Ishida H, Takeuchi Y, Kashida H, Kiriyama S, Hori S, Lee K, Tashiro J, Kobayashi N, Nakajima T, Suzuki S, Mutoh M; J-FAPP Study III Group. Intensive endoscopic resection for downstaging of polyp burden in patients with familial adenomatous polyposis (J-FAPP Study III): a multicenter prospective interventional study. Endoscopy. 2023 Apr;55(4):344-352. doi: 10.1055/a-1945-9120. Epub 2022 Oct 10. PMID 36216266
- [Derived] Motz VL, Lester C, Moyer MT, Maranki JL, Levenick JM. Hybrid argon plasma coagulation-assisted endoscopic mucosal resection for large sessile colon polyps to reduce local recurrence: a prospective pilot study. Endoscopy. 2022 Jun;54(6):580-584. doi: 10.1055/a-1677-3954. Epub 2021 Dec 14. PMID 34905795
- [Derived] Park E, Barge W, Kramer J, Alajati B, Jakate S, Cimbaluk D, Giusto D, Ritz E, Bishehsari F, Lee S, Singh S, Losurdo J, Brown M, DeMeo M, Abraham R, Ma K, Melson J. Interobserver reliability of methods to determine complete resection of adenomas in colonoscopy. Endoscopy. 2021 Dec;53(12):1250-1255. doi: 10.1055/a-1331-4446. Epub 2021 Feb 18. PMID 33285582
- [Derived] de Benito Sanz M, Hernandez L, Garcia Martinez MI, Diez-Redondo P, Joao Matias D, Gonzalez-Santiago JM, Ibanez M, Nunez Rodriguez MH, Cimavilla M, Tafur C, Mata L, Guardiola-Arevalo A, Feito J, Garcia-Alonso FJ; POLIPEC HOT-COLD Study Group. Efficacy and safety of cold versus hot snare polypectomy for small (5-9 mm) colorectal polyps: a multicenter randomized controlled trial. Endoscopy. 2022 Jan;54(1):35-44. doi: 10.1055/a-1327-8357. Epub 2021 Feb 18. PMID 33264811
- [Derived] Nakamura M, Yano T, Esaki M, Oka S, Mitsui K, Hirai F, Kawasaki K, Fujishiro M, Torisu T, Tanaka S, Iwakiri K, Kishi M, Matsumoto T, Yamamoto H. Novel ultrathin double-balloon endoscopy for the diagnosis of small-bowel diseases: a multicenter nonrandomized study. Endoscopy. 2021 Aug;53(8):802-814. doi: 10.1055/a-1243-0226. Epub 2020 Sep 9. PMID 32906162
- [Derived] Meng W, Yue P, Leung JW, Wang H, Wang X, Wang F, Zhu K, Zhang L, Zhu X, Wang Z, Zhang H, Zhou W, Li X. Impact of mechanical simulator practice on clinical ERCP performance by novice surgical trainees: a randomized controlled trial. Endoscopy. 2020 Nov;52(11):1004-1013. doi: 10.1055/a-1217-6727. Epub 2020 Aug 31. PMID 32869230
- [Derived] Kovacevic B, Klausen P, Rift CV, Toxvaerd A, Grossjohann H, Karstensen JG, Brink L, Hassan H, Kalaitzakis E, Storkholm J, Hansen CP, Hasselby JP, Vilmann P. Clinical impact of endoscopic ultrasound-guided through-the-needle microbiopsy in patients with pancreatic cysts. Endoscopy. 2021 Jan;53(1):44-52. doi: 10.1055/a-1214-6043. Epub 2020 Jul 21. PMID 32693411
- [Derived] Subramaniam S, Kandiah K, Chedgy F, Fogg C, Thayalasekaran S, Alkandari A, Baker-Moffatt M, Dash J, Lyons-Amos M, Longcroft-Wheaton G, Brown J, Bhandari P. A novel self-assembling peptide for hemostasis during endoscopic submucosal dissection: a randomized controlled trial. Endoscopy. 2021 Jan;53(1):27-35. doi: 10.1055/a-1198-0558. Epub 2020 Jul 17. PMID 32679602
- [Derived] Zhang Y, Liu L, Wang Q, Guo L, Ye L, Zeng H, Zeng X, Yuan X, Li Y, Zhang Y, Zhou E, Hu B. Endoscopic submucosal dissection with additional radiotherapy in the treatment of T1a esophageal squamous cell cancer: randomized controlled Trial. Endoscopy. 2020 Dec;52(12):1066-1074. doi: 10.1055/a-1198-5232. Epub 2020 Jul 15. PMID 32668474
- [Derived] Seicean A, Samarghitan A, Bolboaca SD, Pojoga C, Rusu I, Rusu D, Sparchez Z, Gheorghiu M, Al Hajjar N, Seicean R. Contrast-enhanced harmonic versus standard endoscopic ultrasound-guided fine-needle aspiration in solid pancreatic lesions: a single-center prospective randomized trial. Endoscopy. 2020 Dec;52(12):1084-1090. doi: 10.1055/a-1193-4954. Epub 2020 Jul 10. PMID 32650346
- [Derived] Alvarez-Gonzalez MA, Pantaleon Sanchez MA, Bernad Cabredo B, Garcia-Rodriguez A, Frago Larramona S, Nogales O, Diez Redondo P, Puig Del Castillo I, Romero Mascarell C, Caballero N, Romero Sanchez-Miguel I, Perez Berbegal R, Hernandez Negrin D, Bujedo Sadornill G, Perez Oltra A, Casals Urquiza G, Amoros Martinez J, Seoane Urgorri A, Ibanez Zafon IA, Gimeno-Garcia AZ. Educational nurse-led telephone intervention shortly before colonoscopy as a salvage strategy after previous bowel preparation failure: a multicenter randomized trial. Endoscopy. 2020 Nov;52(11):1026-1035. doi: 10.1055/a-1178-9844. Epub 2020 Jun 17. PMID 32557475
- [Derived] Struyvenberg M, Kahn A, Fleischer D, Swager AF, Bouma B, Ganguly EK, Konda V, Lightdale CJ, Pleskow D, Sethi A, Smith M, Trindade AJ, Wallace MB, Wang K, Wolfsen HC, Tearney GJ, Curvers WL, Leggett CL, Bergman JJ. Expert assessment on volumetric laser endomicroscopy full scans in Barrett's esophagus patients with or without high grade dysplasia or early cancer. Endoscopy. 2021 Mar;53(3):218-225. doi: 10.1055/a-1194-0397. Epub 2020 Jun 17. PMID 32515006
- [Derived] Zwager LW, Bastiaansen BAJ, Bronzwaer MES, van der Spek BW, Heine GDN, Haasnoot KJC, van der Sluis H, Perk LE, Boonstra JJ, Rietdijk ST, Wolters HJ, Weusten BLAM, Gilissen LPL, Ten Hove WR, Nagengast WB, Bekkering FC, Schwartz MP, Terhaar Sive Droste JS, Vlug MS, Houben MHMG, Rando Munoz FJ, Seerden TCJ, Beaumont H, de Ridder R, Dekker E, Fockens P; Dutch eFTR Group. Endoscopic full-thickness resection (eFTR) of colorectal lesions: results from the Dutch colorectal eFTR registry. Endoscopy. 2020 Nov;52(11):1014-1023. doi: 10.1055/a-1176-1107. Epub 2020 Jun 4. PMID 32498100
- [Derived] Karsenti D, Palazzo L, Perrot B, Zago J, Lemaistre AI, Cros J, Napoleon B. 22G Acquire vs. 20G Procore needle for endoscopic ultrasound-guided biopsy of pancreatic masses: a randomized study comparing histologic sample quantity and diagnostic accuracy. Endoscopy. 2020 Sep;52(9):747-753. doi: 10.1055/a-1160-5485. Epub 2020 May 14. PMID 32408361